CLINICAL TRIAL: NCT01855412
Title: LIBERTY 360: Prospective, Observational, Multi-Center Clinical Study to Evaluate Acute and Long Term Clinical and Economic Outcomes of Endovascular Device Intervention in Patients With Distal Outflow Peripheral Arterial Disease (PAD)
Brief Title: Observational Study to Evaluate PAD Treatment Clinical and Economic Outcomes
Acronym: LIBERTY
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN-0001-P
Record Dates: First submitted 2013-05-07; First posted 2013-05-16 (Estimated); Results first posted 2021-05-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Peripheral Arterial Occlusive Disease
Keywords: PAD; LIBERTY; Observational
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Claudication (Rutherford 2-3): Patients who have been diagnosed with PAD and are classified as on the Rutherford Scale as Rutherford 2-3. Patients may be treated with any FDA-cleared endovascular PAD treatment.
  Interventions: Other: PAD endovascular treatments
- CLI Rutherford 4-5: Patients who have been diagnosed with PAD and classified on the Rutherford Scale as Rutherford 4-5. Patients may be treated with any FDA-cleared endovascular PAD treatment.
  Interventions: Other: PAD endovascular treatments
- CLI Rutherford 6: Patients who have been diagnosed with PAD and classified on the Rutherford Scale as Rutherford 6. Patients may be treated with any FDA-cleared endovascular PAD treatment.
  Interventions: Other: PAD endovascular treatments

INTERVENTIONS:
Other: PAD endovascular treatments — All FDA-cleared endovascular PAD treatments

SUMMARY:
The purpose of this study is to evaluate acute and long term clinical and economic outcomes of endovascular procedures to treat Peripheral Arterial Disease (PAD).

DETAILED DESCRIPTION:
This is a prospective, observational, multi-center, clinical study examining predictors of clinical outcomes for patients undergoing endovascular treatment of lesions within or extending into the target area (10 cm above the medial epicondyle to the digital arteries). This includes disease in a vessel located within or extending into the distal superficial femoral artery (SFA), popliteal (POP), tibial peroneal trunk (TPT), anterior tibial (AT), posterior tibial (PT), and peroneal tibial (PR) arteries.

ELIGIBILITY:
Inclusion Criteria:

1. Subject's age ≥ 18 years.
2. Subject presents with a Rutherford classification of 2 to 6.
3. Subject presents with clinical evidence of PAD requiring endovascular intervention on one or both limbs that includes a target lesion in a native vessel located within or extending into 10 cm above the medial epicondyle to the digital arteries.

   * If subject presents with bilateral disease, the first limb treated with a lesion in the target area will be considered the target limb.
   * For subjects with one or more wounds on the target limb, the target lesion(s) should be considered the lesion(s) in the vessel(s) that provide(s) blood flow to the wound(s).
4. Subject has at least one lesion in a native vessel located within or extending into the target area that is crossed and treated with an endovascular device.

Exclusion Criteria:

1. Subject is unwilling or unable to sign the IRB-approved informed consent form (ICF).
2. Subject is unable to understand or comply with the study protocol requirements.
3. Subject is currently participating in an investigational drug or other device study that can clinically interfere with the endpoints of this study.
4. Subject requires a conversion from endovascular intervention to a surgical bypass graft for any lesion(s) in the target area, as determined by the Investigator.
5. Subject has an in-stent restenosis in the target area, and this lesion is the only one requiring treatment.
6. Subject is pregnant or planning to become pregnant within the study period.
7. Subject has an anticipated life span of less than one (1) year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been determined by their physician to require endovascular device treatment for their PAD.
Sampling Method: Non-Probability Sample
Enrollment: 1204 (Actual)
Dates: Start 2013-05; Primary Completion 2019-04-11 (Actual); Study Completion 2019-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Gray, MD, Principal Investigator — Columbia University; Gary Ansel, MD, Principal Investigator — Ohio Health; George Adams, MD, Principal Investigator — Rex Healthcare; Jihad Mustapha, MD, Principal Investigator — Advanced Cardiac & Vascular Centers
Locations (52):
- United States (52):
  - Mercy Gilbert Medical Center, Gilbert, Arizona
  - Phoenix Heart Cardiovascular, Glendale, Arizona
  - St. Luke's Medical Center, Phoenix, Arizona
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Cedars-Sinai Heart Institute, Los Angeles, California
  - Denver Heart, Denver, Colorado
  - VA Eastern Colorado Healthcare System, Denver, Colorado
  - Colorado Heart and Vascular, PC, Lakewood, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Clearwater Cardiovascular Consultants, Clearwater, Florida
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Lakeland Regional Medical Center, Lakeland, Florida
  - The Heart Institute of Largo, Largo, Florida
  - Baptist Cardiac and Vascular Institute, Miami, Florida
  - Mount Sinai Medical Center Heart Institute, Miami Beach, Florida
  - Florida Hospital, Orlando, Florida
  - Coastal Vascular and Intervention, Pensacola, Florida
  - Pepin Heart Institute, Tampa, Florida
  - Memorial Hospital Carbondale, Carbondale, Illinois
  - Chicago Vascular Clinic, Schaumburg, Illinois
  - St. John's Hospital Springfield, Springfield, Illinois
  - Midwest Cardiovascular Research Foundation, Davenport, Iowa
  - St. Joseph Hospital, Lexington, Kentucky
  - Shady Grove Adventist Hospital, Rockville, Maryland
  - Michigan Outpatient Vascular Institute, Dearborn, Michigan
  - St. John Hospital and Medical Center, Detroit, Michigan
  - Mid-Michigan Heart and Vascular Center, Saginaw, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Metropolitan Heart and Vascular Institute, Coon Rapids, Minnesota
  - Stern Cardiovascular Foundation, Southaven, Mississippi
  - St. Luke's Hospital, Kansas City, Missouri
  - Cox Health System, Springfield, Missouri
  - Gotham Cardiovascular Research, New York, New York
  - Columbia University Medical Center, New York, New York
  - Duke University Hospital, Lumberton, North Carolina
  - Rex Heathcare, Raleigh, North Carolina
  - Ohio Health, Columbus, Ohio
  - St. John Health System, Tulsa, Oklahoma
  - Sanford Research, Sioux Falls, South Dakota
  - University Surgical Associates, Chattanooga, Tennessee
  - Wellmont CVA Heart Institute, Kingsport, Tennessee
  - Premier Surgical Associates, Knoxville, Tennessee
  - Cardiothoracic and Vascular Surgeons, P.A., Austin, Texas
  - El Paso Cardiology Associates, El Paso, Texas
  - University of Texas Medical Branch at Galveston, Galveston, Texas
  - Houston Methodist Research Institute, Houston, Texas
  - Mission Research Institute, New Braunfels, Texas
  - San Antonio Endovascular & Heart Institute, San Antonio, Texas
  - Houston Methodist Research Institute Sugar Land, Sugar Land, Texas
  - Cardiovascular Associates of East Texas, Tyler, Texas
  - Providence Health Services, Waco, Texas

REFERENCES:
- [Background] Adams GL, Mustapha J, Gray W, Hargus NJ, Martinsen BJ, Ansel G, Jaff MR. The LIBERTY study: Design of a prospective, observational, multicenter trial to evaluate the acute and long-term clinical and economic outcomes of real-world endovascular device interventions in treating peripheral artery disease. Am Heart J. 2016 Apr;174:14-21. doi: 10.1016/j.ahj.2015.12.013. Epub 2015 Dec 30. PMID 26995365
- [Result] Mustapha J, Gray W, Martinsen BJ, Bolduan RW, Adams GL, Ansel G, Jaff MR. One-Year Results of the LIBERTY 360 Study: Evaluation of Acute and Midterm Clinical Outcomes of Peripheral Endovascular Device Interventions. J Endovasc Ther. 2019 Apr;26(2):143-154. doi: 10.1177/1526602819827295. Epub 2019 Feb 6. PMID 30722718
- [Result] Mustapha JA, Igyarto Z, O'Connor D, Armstrong EJ, Iorio AR, Driver VR, Saab F, Behrens AN, Martinsen BJ, Adams GL. One-Year Outcomes of Peripheral Endovascular Device Intervention in Critical Limb Ischemia Patients: Sub-Analysis of the LIBERTY 360 Study. Vasc Health Risk Manag. 2020 Feb 10;16:57-66. doi: 10.2147/VHRM.S230934. eCollection 2020. PMID 32103970
- [Result] Giannopoulos S, Secemsky EA, Mustapha JA, Adams G, Beasley RE, Pliagas G, Armstrong EJ. Three-Year Outcomes of Orbital Atherectomy for the Endovascular Treatment of Infrainguinal Claudication or Chronic Limb-Threatening Ischemia. J Endovasc Ther. 2020 Oct;27(5):714-725. doi: 10.1177/1526602820935611. Epub 2020 Jul 3. PMID 32618486
- [Result] Giannopoulos S, Shammas NW, Cawich I, Staniloae CS, Adams GL, Armstrong EJ. Sex-Related Differences in the Outcomes of Endovascular Interventions for Chronic Limb-Threatening Ischemia: Results from the LIBERTY 360 Study. Vasc Health Risk Manag. 2020 Jul 8;16:271-284. doi: 10.2147/VHRM.S246528. eCollection 2020. PMID 32753875
- [Result] Narcisse DI, Weissler EH, Rymer JA, Armstrong EJ, Secemsky EA, Gray WA, Mustapha JA, Adams GL, Ansel GM, Patel MR, Jones WS. The impact of chronic kidney disease on outcomes following peripheral vascular intervention. Clin Cardiol. 2020 Nov;43(11):1308-1316. doi: 10.1002/clc.23444. Epub 2020 Aug 11. PMID 32780436
- [Result] Giannopoulos S, Mustapha J, Gray WA, Ansel G, Adams G, Secemsky EA, Armstrong EJ. Three-Year Outcomes From the LIBERTY 360 Study of Endovascular Interventions for Peripheral Artery Disease Stratified by Rutherford Category. J Endovasc Ther. 2021 Apr;28(2):262-274. doi: 10.1177/1526602820962972. Epub 2020 Oct 5. PMID 33016805
- [Result] Weissler EH, Narcisse DI, Rymer JA, Armstrong EJ, Secemsky E, Gray WA, Mustapha JA, Adams GL, Ansel GM, Patel MR, Jones WS. Characteristics and Outcomes of Patients With Diabetes Mellitus Undergoing Peripheral Vascular Intervention for Infrainguinal Symptomatic Peripheral Artery Disease. Vasc Endovascular Surg. 2021 Feb;55(2):124-134. doi: 10.1177/1538574420968671. Epub 2020 Oct 23. PMID 33094679
- [Result] Magnuson EA, Li H, Vilain K, Armstrong EJ, Secemsky EA, Giannopoulos S, Adams GL, Mustapha J, Cohen DJ; LIBERTY 360 degrees Trial Investigators. Two-year PAD-related health care costs in patients undergoing lower extremity endovascular revascularization: results from the LIBERTY 360 degrees trial. J Med Econ. 2021 Jan-Dec;24(1):570-580. doi: 10.1080/13696998.2021.1917141. PMID 33866936
- [Result] Giannopoulos S, Pliagas G, Armstrong EJ. Procedural and 3-Year Outcomes of Peripheral Vascular Interventions Performed in Office-Based Labs: LIBERTY 360 Sub-Analysis. J Invasive Cardiol. 2021 May;33(5):E365-E377. doi: 10.25270/jic/20.00594. PMID 33932282
- [Result] Giannopoulos, S, Fakorede FA, Cawich I, Dishmon D, Horne A, Raja ML, Mustapha JA, Adams GL, Armstrong EJ. Racial Disparities in Risk for Major Amputation or Death After Endovascular Interventions for Peripheral Artery Disease: A LIBERTY 360 Study. J Crit Limb Ischemia. 2021 June;1(2):E62-E72.
- [Result] Salahuddin T, Giannopoulos S, Adams G, Armstrong EJ. Anterior, posterior, or all-vessel infrapopliteal revascularization in patients with moderate-severe claudication: Insights from the LIBERTY 360 study. Catheter Cardiovasc Interv. 2021 Sep;98(3):559-569. doi: 10.1002/ccd.29780. Epub 2021 May 31. PMID 34057276
- [Result] Jammeh ML, Suggs J, Adams GL, Armstrong EJ, Mustapha J, Zayed MA. Outcomes of Orbital Atherectomy in Patients with Critical Limb Threatening Ischemia and Diabetes. J Crit Limb Ischemia. 2022 Jun;2(2):E29-E37. Epub 2022 Apr 12. PMID 37066103
- [Result] Metser G, Puma J, Mustapha J, Adams GL, Ratcliffe J, Khullar P, Rosero JHC, Armstrong EJ, Zayed M, Green P. Clinical Outcomes of Additional Below-The-Ankle Intervention Compared to Below-The-Knee Intervention Alone: A Post-Hoc Analysis of a Prospective Multicenter Study. J Endovasc Ther. 2023 Oct;30(5):711-720. doi: 10.1177/15266028221092981. Epub 2022 May 3. PMID 35503774

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A subject was considered enrolled when a signed informed consent was in place and all inclusion/no exclusion criteria were met.
Groups:
- Claudication (Rutherford 2-3): Patients who have been diagnosed with PAD and are classified on the Rutherford Scale as Rutherford 2-3.
  PAD endovascular treatments: Patients may be treated with any approved or cleared FDA endovascular devices, per physician choice.
- CLI Rutherford 4-5: Patients who have been diagnosed with PAD and are classified on the Rutherford Scale as Rutherford 4-5.
  PAD endovascular treatments: Patients may be treated with any approved or cleared FDA endovascular devices, per physician choice.
- CLI Rutherford 6: Patients who have been diagnosed with PAD and are classified on the Rutherford Scale as Rutherford 6.
  PAD endovascular treatments: Patients may be treated with any approved or cleared FDA endovascular devices, per physician choice.
Period: Overall Study
Arm/Group | Claudication (Rutherford 2-3) | CLI Rutherford 4-5 | CLI Rutherford 6
Started | 501 | 603 | 100
Completed | 289 | 260 | 24
Not Completed | 212 | 343 | 76
Not completed — Death | 77 | 123 | 30
Not completed — Lost to Follow-up | 28 | 46 | 15
Not completed — Withdrawal by Subject | 77 | 123 | 24
Not completed — Physician Decision | 25 | 31 | 3
Not completed — Site Closure | 4 | 18 | 1
Not completed — Reason not Specified | 1 | 2 | 3

BASELINE CHARACTERISTICS:
Population: Baseline analysis population consists of data from 1,189 enrolled subjects with Investigator signed baseline and procedure patient records. Due to site closure and lack of Investigator signature, 15 subjects were excluded from the cohort.
Groups:
- Total: Total of all reporting groups
Arm/Group | Claudication (Rutherford 2-3) | CLI Rutherford 4-5 | CLI Rutherford 6 | Total
Number analyzed (Participants) | 500 | 589 | 100 | 1189
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age was not collected for one subject in the CLI Rutherford 6 group.
  years
    number analyzed (Participants) | 500 | 589 | 99 | 1188
    (all) | 69.7 (10.0) | 70.3 (10.9) | 68.0 (13.0) | 69.8 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 167 | 225 | 27 | 419
  Male | 333 | 364 | 73 | 770
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 77 | 63 | 29 | 169
  Not Hispanic or Latino | 423 | 526 | 71 | 1020
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 411 | 483 | 78 | 972
  Black or African American | 68 | 89 | 21 | 178
  Asian | 5 | 1 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 2
  Native American | 1 | 4 | 0 | 5
  Other | 14 | 11 | 0 | 25
Region of Enrollment [Number; unit: participants]
  United States | 500 | 589 | 100 | 1189
Baseline Rutherford Classification (RC) [Count of Participants; unit: Participants] — Rutherford Classification (RC) is a commonly used clinical grading system for describing peripheral arterial disease (PAD) on a scale of 0 to 6. RC 6 is the most severe form of PAD.
  There are seven Rutherford categories used to grade the severity of peripheral artery disease; 0: asymptomatic, 1: mild claudication, 2: moderate claudication, 3: severe claudication, 4: ischemic rest pain, 5: minor tissue loss, 6: major tissue loss.
  Participants
    RC 2 | 97 | 0 | 0 | 97
    RC 3 | 403 | 0 | 0 | 403
    RC 4 | 0 | 285 | 0 | 285
    RC 5 | 0 | 304 | 0 | 304
    RC 6 | 0 | 0 | 100 | 100

OUTCOME MEASURES:

1. Primary Outcome: Procedural Success of Endovascular PAD Treatment(s)
Description: Final post-procedural result of <50% residual stenosis for all treated lesions for a participant during index procedure and without angiographic complications as determined by the Angiographic Core Laboratory.
Time Frame: Participants were followed from baseline procedure through hospital discharge, an expected average of less than 24 hours
Population: Analysis population consists of data from 1,106 enrolled subjects with sufficient information to assess procedural success. Fifteen subjects were excluded due to site closure and lack of investigator signature, 83 subjects were excluded due to lack of sufficient stenosis and/or angiographic complication data to determine success or failure.
Measure: Number (95% Confidence Interval); unit: percent of procedures
Arm/Group | Claudication (Rutherford 2-3) | CLI Rutherford 4-5 | CLI Rutherford 6
Number analyzed (Participants) | 469 | 545 | 92
percent of procedures | 83.6 [79.9 to 86.8] | 75.8 [72.0 to 79.3] | 68.5 [58.0 to 77.8]

2. Primary Outcome: Lesion Success of Endovascular PAD Treatment(s)
Description: Final post-procedural result of <50% residual stenosis for a given lesion treated during index procedure without angiographic complications as determined by the Angiographic Core Laboratory.
Time Frame: as for outcome 1
Population: Analysis population consists of data from 1,452 treated lesions with sufficient information to assess procedural success. Data from fifteen subjects were excluded due to site closure and lack of investigator signature; 76 lesions were excluded due to lack of sufficient stenosis and/or angiographic complication data to determine success or failure.
Measure: Number (95% Confidence Interval); unit: percent of lesions treated
Arm/Group | Claudication (Rutherford 2-3) | CLI Rutherford 4-5 | CLI Rutherford 6
Number analyzed (Participants) | 578 | 733 | 141
percent of lesions treated | 84.9 [81.9 to 88.0] | 79.1 [75.8 to 82.1] | 75.2 [66.8 to 82.2]

3. Primary Outcome: Rate of Freedom From Major Adverse Events (MAEs) at One (1) and Three (3) Years
Description: A Kaplan-Meier analysis was performed to determine the percent probability that the study participant was free from a major adverse event through 1 year and 3 years.
  1- and 3-year MAE is composed of:
  * Death within 30 days of index procedure
  * Unplanned major (above the ankle) amputation of the target limb
  * Clinically-driven TVR (Target Vessel Revascularization) of the target limb
Time Frame: One (1) year and three (3) years post-procedure
Population: Analysis population consists of data from 1,189 enrolled subjects with Investigator signed baseline and procedure patient records. Due to site closure and lack of Investigator signature, 15 subjects were excluded in the cohort.
Measure: Number (95% Confidence Interval); unit: percent probability of freedom from MAE
Arm/Group | Claudication (Rutherford 2-3) | CLI Rutherford 4-5 | CLI Rutherford 6
Number analyzed (Participants) | 500 | 589 | 100
percent probability of freedom from MAE
  Freedom from MAE at 1-Year | 82.1 [78.6 to 85.7] | 73.2 [69.4 to 77.0] | 59.3 [48.4 to 70.1]
  Freedom from MAE at 3-Years | 70.3 [65.9 to 74.7] | 62.0 [57.5 to 66.5] | 47.4 [34.7 to 60.0]

ADVERSE EVENTS:
Time Frame: Index procedure through 5 years
Groups:
- Claudication Rutherford 2-3 Procedure Through 30 Days: Patients who have been diagnosed with PAD and are classified on the Rutherford Scale as Rutherford 2-3.
  PAD endovascular treatments: Patients may be treated with any approved or cleared FDA endovascular devices, per physician choice.
- CLI Rutherford 4-5 Procedure Through 30 Days: Patients who have been diagnosed with PAD and are classified on the Rutherford Scale as Rutherford 4-5.
  PAD endovascular treatments: Patients may be treated with any approved or cleared FDA endovascular devices, per physician choice.
- CLI Rutherford 6 Procedure Through 30 Days: Patients who have been diagnosed with PAD and are classified on the Rutherford Scale as Rutherford 6.
  PAD endovascular treatments: Patients may be treated with any approved or cleared FDA endovascular devices, per physician choice.
- Rutherford 2-3 31 Days - 365 Days Post-Procedure: Patients who have been diagnosed with PAD and are classified on the Rutherford Scale as Rutherford 2-3.
  PAD endovascular treatments: Patients may be treated with any approved or cleared FDA endovascular devices, per physician choice.
  Adverse events occurring between 31 Days - 365 Days Post-Procedure
- CLI Rutherford 4-5 31 Days - 365 Days Post-Procedure: Patients who have been diagnosed with PAD and are classified on the Rutherford Scale as Rutherford 4-5.
  PAD endovascular treatments: Patients may be treated with any approved or cleared FDA endovascular devices, per physician choice.
  Adverse events occurring between 31 Days - 365 Days Post-Procedure
- CLI Rutherford 6 31 Days - 365 Days Post-Procedure: Patients who have been diagnosed with PAD and are classified on the Rutherford Scale as Rutherford 6.
  PAD endovascular treatments: Patients may be treated with any approved or cleared FDA endovascular devices, per physician choice.
  Adverse events occurring between 31 Days - 365 Days Post-Procedure
- Claudication Rutherford 2-3 366 Days Post-Procedure or Greater: Patients who have been diagnosed with PAD and are classified on the Rutherford Scale as Rutherford 2-3.
  PAD endovascular treatments: Patients may be treated with any approved or cleared FDA endovascular devices, per physician choice.
  Adverse events occurring between 366 Days Post-Procedure or Greater
- CLI Rutherford 4-5 366 Days Post-Procedure or Greater: Patients who have been diagnosed with PAD and are classified on the Rutherford Scale as Rutherford 4-5.
  PAD endovascular treatments: Patients may be treated with any approved or cleared FDA endovascular devices, per physician choice.
  Adverse events occurring between 366 Days Post-Procedure or Greater
- CLI Rutherford 6 366 Days Post-Procedure or Greater: Patients who have been diagnosed with PAD and are classified on the Rutherford Scale as Rutherford 6.
  PAD endovascular treatments: Patients may be treated with any approved or cleared FDA endovascular devices, per physician choice.
  Adverse events occurring between 366 Days Post-Procedure or Greater
Arm/Group | Claudication Rutherford 2-3 Procedure Through 30 Days | CLI Rutherford 4-5 Procedure Through 30 Days | CLI Rutherford 6 Procedure Through 30 Days | Rutherford 2-3 31 Days - 365 Days Post-Procedure | CLI Rutherford 4-5 31 Days - 365 Days Post-Procedure | CLI Rutherford 6 31 Days - 365 Days Post-Procedure | Claudication Rutherford 2-3 366 Days Post-Procedure or Greater | CLI Rutherford 4-5 366 Days Post-Procedure or Greater | CLI Rutherford 6 366 Days Post-Procedure or Greater
All-Cause Mortality (participants affected / at risk) | 2/501 | 2/603 | 4/100 | 18/501 | 40/603 | 17/100 | 57/501 | 81/603 | 9/100
Serious Adverse Events (participants affected / at risk) | 72/501 | 112/603 | 24/100 | 145/501 | 249/603 | 40/100 | 167/501 | 227/603 | 24/100
Other Adverse Events (participants affected / at risk) | 28/501 | 31/603 | 2/100 | 0/501 | 0/603 | 0/100 | 0/501 | 0/603 | 0/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Claudication Rutherford 2-3 Procedure Through 30 Days (N=501) | CLI Rutherford 4-5 Procedure Through 30 Days (N=603) | CLI Rutherford 6 Procedure Through 30 Days (N=100) | Rutherford 2-3 31 Days - 365 Days Post-Procedure (N=501) | CLI Rutherford 4-5 31 Days - 365 Days Post-Procedure (N=603) | CLI Rutherford 6 31 Days - 365 Days Post-Procedure (N=100) | Claudication Rutherford 2-3 366 Days Post-Procedure or Greater (N=501) | CLI Rutherford 4-5 366 Days Post-Procedure or Greater (N=603) | CLI Rutherford 6 366 Days Post-Procedure or Greater (N=100)
Arrhythmias (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Cardiac dysfunction - Chronic heart failure or aggravated (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Cardiac/cardiopulmonary arrest (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 4 (4) | 1 (1) | 4 (4) | 9 (9) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Coronary artery thrombus/thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 6 (6) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 2 (2) | 4 (4) | 0 (0)
Other cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Gastrointestional infection/inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Other digestive disorders (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergic reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood and lymphatic system disorder-anemia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 6 (6) | 0 (0)
Compartment syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death-unknown cause (General disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 10 (10) | 7 (7) | 19 (19) | 23 (23) | 4 (4)
Infection-Systemic (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 1 (1) | 2 (2) | 4 (4) | 0 (0)
Injury/trauma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 4 (4) | 5 (5) | 1 (1)
Other adverse event (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Shock (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Hepatic-biliary system disorders (e.g. liver, bile duct) (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Other peripheral procedural complication (Injury, poisoning and procedural complications) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral arteriovenous fistula (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery abrupt closure (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery dissection (Injury, poisoning and procedural complications) | 43 (46) | 28 (30) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery distal embolization (Injury, poisoning and procedural complications) | 3 (3) | 5 (7) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery no reflow (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery perforation (Injury, poisoning and procedural complications) | 7 (7) | 7 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery slow flow (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery thrombus/thrombosis (Injury, poisoning and procedural complications) | 6 (6) | 11 (11) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery vasospasm (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (CVA) (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Other neuro/pshychiatric disorders (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Transient ischemic attack (TIA) (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic renal failure or worsened (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 2 (2) | 6 (6) | 0 (0)
Chronic obstructive pulmonary disease (COPD) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bleeding/hemorrhage non-access site (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bleeding/hemorrhage, access site (Vascular disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bruising/hematoma access site (Vascular disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism, pulmonary (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
New/worsening infection (Vascular disorders) | 0 (0) | 8 (8) | 6 (6) | 1 (1) | 27 (30) | 9 (9) | 4 (6) | 17 (17) | 4 (6)
New/worsening pain (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (2) | 3 (3) | 0 (0)
New/worsening wound (Vascular disorders) | 0 (0) | 11 (12) | 10 (11) | 5 (6) | 21 (24) | 11 (14) | 9 (11) | 15 (21) | 2 (2)
Other peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Other vascular disorder (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Peripheral artery restenosis (Vascular disorders) | 1 (1) | 15 (17) | 2 (2) | 80 (107) | 131 (212) | 18 (23) | 85 (160) | 130 (326) | 10 (17)
Peripheral artery stenosis (Vascular disorders) | 6 (6) | 18 (20) | 2 (2) | 71 (89) | 129 (164) | 11 (11) | 76 (102) | 95 (132) | 4 (5)
Peripheral artery/vascular disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Peripheral thrombus/thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Claudication Rutherford 2-3 Procedure Through 30 Days (N=501) | CLI Rutherford 4-5 Procedure Through 30 Days (N=603) | CLI Rutherford 6 Procedure Through 30 Days (N=100) | Rutherford 2-3 31 Days - 365 Days Post-Procedure (N=501) | CLI Rutherford 4-5 31 Days - 365 Days Post-Procedure (N=603) | CLI Rutherford 6 31 Days - 365 Days Post-Procedure (N=100) | Claudication Rutherford 2-3 366 Days Post-Procedure or Greater (N=501) | CLI Rutherford 4-5 366 Days Post-Procedure or Greater (N=603) | CLI Rutherford 6 366 Days Post-Procedure or Greater (N=100)
Peripheral artery dissection (Injury, poisoning and procedural complications) | 28 (29) | 31 (35) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2014-08-21): https://cdn.clinicaltrials.gov/large-docs/12/NCT01855412/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-24): https://cdn.clinicaltrials.gov/large-docs/12/NCT01855412/SAP_001.pdf